CLINICAL TRIAL: NCT04794465
Title: Asymptomatic Inflammatory Bowel Disease Diagnosed During the Colorectal Cancer Population Screening un Catalonia
Brief Title: Asymptomatic Inflammatory Bowel Disease in Catalonia
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Anna Selva, Clinical Epidemiology and Cancer Screening, Corporació Sanitària Parc Taulí, Sabadell, Spain, Corporacion Parc Tauli
Other Study IDs: 2021/5006
Record Dates: First submitted 2021-03-07; First posted 2021-03-12 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Inflammatory Bowel Diseases
Keywords: inflammatory bowel disease; epidemiology
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Asymptomatic IBD diagnosed during the colorectal cancer screening
  Interventions: Diagnostic Test: Colorectal cancer screening

INTERVENTIONS:
Diagnostic Test: Colorectal cancer screening — Patients with IBP diagnosed during the colorectal cancer screening

SUMMARY:
An early treatment of inflammatory bowel disease (IBD) has been proposed to correlate to better outcomes. In Catalonia the screening programme was implemented in all the territory in 2015. The aim of this study is to describe the natural history of the asymptomatic IBD detected during colorectal cancer population screening.

DETAILED DESCRIPTION:
This study will be performed and reported according to the STROBE Statement guidelines ( http://www.strobe-statement.org/index.php?id=strobe-home).

Design:

Observational, multicentre and retrospective cohort study.

Centre selection and recruitment:

All the participating centres in population colorectal cancer screening in Catalonia will be invited. All the participating centres must certify the approval of the protocol in their ethical committees.

Study population:

All patients with asymptomatic IBD diagnosed during the population colorectal cancer screening in the Catalonian colorectal screening program within the period 2000 to 2019 will be included.

Study variables

Prevalence of asymptomatic IBD diagnosed and their evolution through the years will be described. The following variables will be collected (annex1):

* Sex (male, female)
* Age
* Fecal immunotest (value)
* Date of screening colonoscopy (yyyy/mm/dd)
* Ileoscopy performed (yes/no)
* Type of IBD (CD, UC, indeterminate colitis)
* Endoscopic findings: mild-moderate activity or severe activity for CD and Mayo score for UC (value of the scores).
* Montreal classification (value of the classification)
* Histology (diagnostic, compatible, unspecific or no compatible)
* Microscopic description (cryptitis, abscess, mucus depletion, granuloma, architectural pattern alteration
* Past medical history, smoking habit, previous abdominal surgeries and comorbidities.
* Familiar history of IBD
* Extraintestinal manifestations (cutaneous, ophthalmologic, articular)
* Other studies performed (endoscopic capsule, MRI, gastroscopy, echography).
* Calprotectin: value of the first analysis in the outpatient visit.
* Blood test: Haemoglobin, ferritin and PCR: values of the first analysis in the outpatient visit.
* Fist symptom: none, change in depositional rhythm, abdominal pain, weight loss, rectal urgency, anal pain, iron deficiency anaemia.
* Date of first IBD symptom (yyyy/mm/dd)
* Time to first IBD symptom: time in days from the diagnosis of IBD.
* Treatments used: none; 5- aminosalicylates, corticosteroids, non-biologic immunosuppressive treatment, biologic treatment, surgery
* Treatment start and end date (yyyy/mm/dd)
* Time to first treatment: time in days from the diagnosis of IBD.
* Follow-up endoscopy: Date (yyyy/mm/dd) and activity.

Data collection:

All patients with asymptomatic IBD diagnosed during the population colorectal cancer screening within the period 2000 to 2019 will be identified by the colorectal cancer screening program registry.

Patient identity will be given to a data manager. This manager will administrate the data of each patient in their hospital.

The person in charge of the study in each hospital will collect the anonymized data using REDCap database (Research Electronic Data Capture), a secure, web-based application designed to support data collection form research studies.

Statistical methods:

Categorical variable will be given as natural frequencies and percentages and quantitative variables will be given as mean or median and standard deviation or interquartile ranges. Kaplan-Meier analysis will be used to describe the time to first symptom and or time to first treatment. If necessary, the long rank test will be used to compare survival curves. A multivariate Cox analysis will be performed to ascertain the independent predictors of aggressive disease.

Ethical issues:

The research will use retrospective anonymized data from the technical screening office of Catalonia. No personal data will be used, and all the patient data will be encrypted, so that no personal identification would be retrievable or traceable to the original source from the working database.

All the researchers who collaborate in the study will sign a commitment document in which their functions and obligations will be defined. Both in the collection of data and in the analysis, Organic Law 3/2018, of December 5, on the Protection of Personal Data and guarantee of digital rights and the provisions of European Regulation 679/2016 will be followed.

The study was revised and approved by the local ethics committee of the Hospital universitarian Parc Tauli in Sabadell (CEIC 2021/5006) on 15 February 2021. The study will comply with the ethical guidelines of the Declaration of Helsinki. Therefore, as the study uses retrospective anonymized data and it has no impact on evolution or treatment patient, there is no need to obtain informed consent. The study will be performed in accordance with the STROBE statement for reporting observational studies in Epidemiology.

ELIGIBILITY:
Inclusion Criteria:

* All patients with asymptomatic IBD diagnosed during the population colorectal cancer screening in the Catalonian colorectal screening program within the period 2000 to 2019 will be included.

Exclusion Criteria:

* Symptoms in the first outpatient visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Centre selection and recruitment:
  All the participating centres in population colorectal cancer screening in Catalonia will be invited. All the participating centres must certify the approval of the protocol in their ethical committees.
  Study population:
  All patients with asymptomatic IBD diagnosed during the population colorectal cancer screening in the Catalonian colorectal screening program within the period 2000 to 2019 will be included.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2021-07-15 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
Time to treatment | From date of diagnosis until the date of first treatment, assessed up to 19 years.
  To see the evolution of the asymptomatic IBD and the need for the treatment

SECONDARY OUTCOMES:
Time to symptoms | From date of diagnosis until the date of first symptom, assessed up to 19 years.
  To see the evolution of the asymptomatic IBD and the symptomatology

CONTACTS AND LOCATIONS:
Locations (1):
- Corporació Sanitària Parc Taulí, Sabadell, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No